CLINICAL TRIAL: NCT00569335
Title: Phase II Trial of Combination Therapy With S-1, Irinotecan, and Bevacizumab (SIRB) in Patients With Unresectable or Recurrent Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01023020
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Colorectal, Cancer
Keywords: S-1, Bevacizumab, Irinotecan
MeSH Terms: conditions — Colonic Neoplasms | interventions — S 1 (combination); Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): S-1, Irinotecan, Bevacizumab
  Interventions: Drug: S-1, Irinotecan, Bevacizumab

INTERVENTIONS:
Drug: S-1, Irinotecan, Bevacizumab — S-1 is administered orally on days 1 to 14 of a 21-day cycle. Patients are assigned on the basis of body surface area (BSA) to receive one of the following oral doses twice daily: 40 mg (BSA <1.25m2), 50 mg (BSA >1.25 to <1.50 m2), or 60 mg (BSA >1.50 m2).
  Irinotecan 150 mg/m2 is administered by intravenous infusion on day 1. Bevacizumab 7.5 mg/kg (body weight) is administered by intravenous infusion on day 1.

SUMMARY:
Phase II trial of combination therapy with S-1, irinotecan, and bevacizumab (SIRB) in patients with unresectable or recurrent colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal carcinoma with inoperable, locally advanced, or metastatic disease, not amenable to curative therapy
2. Measurable disease or non-measurable but assessable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST)
3. Patients with no previous treatment (radiotherapy or chemotherapy). Patients who have received postoperative adjuvant chemotherapy are eligible if relapse is diagnosed more than 180 days after the end of such treatment.

   Preoperative or postoperative irradiation (<30 Gy) for rectal cancer is possible
4. Age >20 years
5. Life expectancy of at least 3 months
6. ECOG PS of 0 or 1
7. Adequate function of major organs as defined below:

   1. Hemoglobin >9.0 g/dL
   2. White blood cell count >3,000/mm3
   3. Neutrophil count >1,500/mm3
   4. Platelet count >100,000/mm3
   5. Total bilirubin <1.5 mg/dL
   6. AST and ALT <100 U/L (<200 U/L in patients with liver metastasis)
   7. Serum creatinine <1.2 mg/dL
   8. Creatinine clearance estimate by the Cockcroft-Gault method >50 mL/min (reduce initial dosage by one step if ≥50 but <80 mL/min)
8. Able to take capsules orally.
9. No electrocardiographic abnormalities within 28 days before enrollment that would clinically preclude the execution of the study, as judged by the investigator.
10. Voluntary written informed consent.

Exclusion Criteria:

1. Serious drug hypersensitivity or a history of drug allergy
2. Active double cancer
3. Active infections (e.g., patients with pyrexia of 38℃ or higher)
4. History of gastrointestinal perforation, intestinal tract paralysis, or ileus within 1 year.
5. Uncontrolled hypertension
6. Serious complications (e.g., pulmonary fibrosis, interstitial pneumonitis, heart failure, renal failure, hepatic failure, or poorly controlled diabetes)
7. Moderate or severe ascites or pleural effusion requiring treatment
8. Watery diarrhea
9. Treatment with flucytosine or atazanavir sulfate
10. Metastasis to the CNS
11. Pregnant women, possibly pregnant women, women wishing to become pregnant, and nursing mothers. Men who are currently attempting to conceive children.
12. Severe mental disorder
13. Continuous treatment with steroids
14. Urine dipstick for proteinuria should be <2+
15. Patient with a past history of thrombosis, cerebral infarction, myocardial infarction, or pulmonary embolism
16. Major surgical procedure, open biopsy, or clinically significant traumatic injury within 4 weeks
17. Long-term daily treatment with aspirin (>325 mg/day)
18. History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
19. Judged ineligible for participation in the study by the investigator for safety reasons.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety | any time

SECONDARY OUTCOMES:
Progression-free survival, Response rate, Overall survival, Time to treatment failure, Treatment situation | every course for first three courses, then every other course

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhide Yamada, Principal Investigator — National Cancer Center Hospital
Locations (1):
- National Cancer Center Hospital, Tsukiji, Chuo-ku, Tokyo, Japan